CLINICAL TRIAL: NCT01981824
Title: Femur Length to Mid-thigh Circumference Ratio in Prediction of IUGR
Brief Title: Prediction of Growth Restricted Fetuses Using Femur Length to Mid-thigh Circumference Ratio: A Case-control Study
Acronym: IUGR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Alaa Sayed Abdul-hafeez, Femur length to mid-thigh circumference ratio in prediction of IUGR, Ain Shams Maternity Hospital
Other Study IDs: 11110000
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-10

CONDITIONS: Fetal Growth Restriction
Keywords: prediction IUGR FL/MTC
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
One of the most challenging areas currently facing obstetricians is the detection and management of pregnancies in which the growth of the fetus is poor. These fetuses have not only increased rates of perinatal morbidity and mortality, but also have higher levels of morbidity extending into adult life (Linda; Murray 2010).

In developing countries including Egypt, low birth weight is a national concern and emphasized in population and health policies according to the latest WHO data published in April 2011 low Birth Weight Deaths in Egypt reached 13,587 or 3.74% of total deaths, Mortality was more frequent in LBW (31.6%) than normal birth weight (NBW) infants (2.0%).

Fetal growth restriction (FGR) is defined as fetuses whose growth velocity slows down or stops completely because of inadequate oxygen and nutritional supply or utilization (Linda; Murray 2010). Low birth weight (LBW) refers to an infant with a birth weight < 2500 g, Small for gestational age (SGA) birth is defined as an estimated fetal weight (EFW) less than the 10th centile and severe SGA as an EFW less than the 3rd centile, (RCOG Green-top Guideline No.31, 2013).

Ultrasound has been used as a tool for determining fetal health and a variety of sonographic parameters have been used to screen and diagnose IUGR including fetal biometry, fetal body proportions (Campbell et al., 1994), amniotic fluid volume (Owen et al., 1999), subcutaneous tissue thickness and estimated fetal weight (EFW) (Larciprete et al., 2005).

IUGR is associated with changes in the body proportions as undernourished fetus directs most of its energy to maintain the growth of vital organs, such as the brain and heart, at the expense of the liver, muscle and fat and this results in decreased abdominal and thigh circumference measurements and hence theoretically increased HC/AC, FL/AC and FL/TC ratios (Colley et al., 1991).

Fetal thigh circumference has a role to play in accurately measuring fetal weight when incorporated with other fetal parameters and provide a potentially straightforward method for assessing the deposition of muscle and fat in the growing fetus; there is a scope of using the FL/TC ratio in predicting IUGR (Sanyal et al., 2012).

Fetal thigh circumference to femur length ratio (FL/TC) seems to be potential for use in predicting IUGR (Shripad; Varalaxmi, 2005).

DETAILED DESCRIPTION:
Aim of work To determine usefulness of antenatally measured femur length to mid thigh circumference ratio to predict intra-uterine growth restricted fetuses.

Study design Observational Case-Control study. Study population This study will be conducted at the department of Obstetrics and Gynecology recruiting pregnant women selected from the attendees of antenatal clinic, emergency department and from inpatient wards of Ain Shams University Maternity Hospital from the period of October 2013 to October 2014.

This study will include 100 pregnant women these cases will divided into 2 groups:

1. Normal growth Fetuses Group: will include 50 pregnant females all in third trimester.
2. IUGR fetuses Group: will include 50 pregnant females all in third trimester.

Inclusion criteria:

1. all pregnant women aged between 20-40 years ,
2. Singleton pregnancy,
3. Gestational age of 28-40 weeks, and
4. Reliable dates by early antenatal ultrasound.

Exclusion criteria:

1. Ultrasonographically detected congenital fetal malformation,
2. Fetal hydrops,
3. Multiple pregnancy,
4. Post-term pregnancy,
5. Intrauterine fetal death.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria:

1. all pregnant women aged between 20-40 years ,
2. Singleton pregnancy,
3. Gestational age of 28-40 weeks, and
4. Reliable dates by early antenatal ultrasound. -

Exclusion Criteria:Exclusion criteria:

1. Ultrasonographically detected congenital fetal malformation,
2. Fetal hydrops,
3. Multiple pregnancy,
4. Post-term pregnancy,
5. Intrauterine fetal death. -

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population This study will be conducted at the department of Obstetrics and Gynecology recruiting pregnant women selected from the attendees of antenatal clinic, emergency department and from inpatient wards of Ain Shams University Maternity Hospital from the period of October 2013 to October 2014.
  This study will include 100 pregnant women these cases will divided into 2 groups:
  1. Normal growth Fetuses Group: will include 50 pregnant females all in third trimester.
  2. IUGR fetuses Group: will include 50 pregnant females all in third trimester.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
femur length to mid-thigh circumference ratio | one year
  To determine usefulness of antenatally measured femur length to mid thigh circumference ratio to predict intra-uterine growth restricted fetuses.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa sayed abdul-Hafeez, MD, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Abbassia, Egypt